CLINICAL TRIAL: NCT02155842
Title: High Versus Moderate Intensity Endurance Exercise Training in Treating Diastolic Heart Failure
Brief Title: Exercise Training in Treating Diastolic Heart Failure
Acronym: TREND-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unforseen problems recruiting patients
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: LHL-Klinikkene, Røros (Other); LHL-Klinikkene, Feiring (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014.12327
Record Dates: First submitted 2014-05-27; First posted 2014-06-04 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure, Diastolic; Ventricular Dysfunction, Left
Keywords: exercise therapy
MeSH Terms: conditions — Heart Failure, Diastolic; Ventricular Dysfunction, Left

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity endurance exercise (Experimental): Four weeks comprehensive cardiac rehabilitation with moderate volume high intensity endurance exercise, followed by 6 months non-supervised endurance exercise
  Interventions: Behavioral: High intensity endurance exercise
- Moderate continuous endurance exercise (Active Comparator): Four weeks comprehensive cardiac rehabilitation with moderate volume moderate intensity endurance exercise, followed by 6 months non-supervised endurance exercise
  Interventions: Behavioral: Moderate continuous endurance exercise

INTERVENTIONS:
Behavioral: High intensity endurance exercise
  Arms: High intensity endurance exercise
Behavioral: Moderate continuous endurance exercise
  Arms: Moderate continuous endurance exercise

SUMMARY:
The purpose of this study is to determine whether endurance exercise of either high or moderate intensity can reverse structural and functional changes of the heart in patients with diastolic heart failure, and to investigate which type of exercise is best in terms of aerobe capacity and quality of life.

The investigators expect that high intensity endurance exercise is superior to moderate intensity endurance exercise.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled intervention study comparing two active arms. Eligible patients are being sampled consecutively by cardiologists, and randomized to either high or moderate intensity endurance exercise. Endpoints are measured at baseline, 4 weeks and 7 months. The intervention is considered safe, and the study has been approved by the Regional Ethics Committee (REK-midt).

This project has been financially supported by the Norwegian ExtraFoundation for Health and Rehabilitation through EXTRA funds.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle
* Normal systolic function left ventricular ejection fraction (LVEF) < 50%
* New York Heart Association (NYHA) class II or III
* Diastolic dysfunction (E/é < 15 or E/é 8-15 and N-terminal proBNP > 220pg/ml)
* Medically stable the last 4 weeks
* Written informed consent

Exclusion Criteria:

* Other causes of dyspnea than diastolic heart failure
* Personal preferences or characteristics prohibiting the person from attending inpatient cardiac rehabilitation
* Not able to perform physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in aerobic capacity measured as oxygen consumption | Baseline and 7 months
  Cardiopulmonary exercise test

SECONDARY OUTCOMES:
Feasibility, measured as attrition rate and compliance with exercise | Baseline to 7 months
Blood-risk profile, measured as changes in cholesterol, hemoglobin, N terminal-proBNP | Baseline to 7 months
Cardiac function measured as volume, size, efficacy | Baseline to 7 months
  Ultrasound
Arterial function measured as blood-vessel elasticity | Baseline to 7 months
  Ultrasound
Quality of life | Baseline to 7 months
  Self-reported questionnaires
Changes in everyday activity level | Baseline to 7 months
  Self-reported questionnaire, diary, activity monitoring device
Change in diastolic filling pressure measured as E/é | Baseline to 7 months
  Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- LHL Klinikkene, Røros, Norway

IPD SHARING:
Plan to Share IPD: No